CLINICAL TRIAL: NCT07200492
Title: Anti-Redness Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ChinaNorm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: C23036010
Record Dates: First submitted 2025-09-11; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Redness
MeSH Terms: conditions — Erythema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Facial Test Arm (Other)
  Interventions: Other: Facial serum application
- Facial Control Arm (No Intervention)
- Arm Test Arm (Other)
  Interventions: Other: Forearm serum application
- Arm Control Arm (No Intervention)

INTERVENTIONS:
Other: Facial serum application — The trained technician will apply the 0.3g-0.4g investigational products on the subject's half face.
  Arms: Facial Test Arm
Other: Forearm serum application — The trained technician will apply the (2mg±0.1mg)/cm² investigational products on the subject's forearm.
  Arms: Arm Test Arm

SUMMARY:
This clinical study is a single-center, randomized, split-face, on-site controlled trial conducted at Shanghai China-Norm Quality Technical Service Co., Ltd. The primary objective is to evaluate the efficacy of Eucerin Ultrasensitive Repair Intensive Source Serum in providing instant and long-lasting (24-hour) soothing and repairing effects under induced redness conditions. The design involves recruiting 30 healthy Chinese female subjects aged 18-60 years, who meet stringent inclusion/exclusion criteria, including absence of skin conditions and no recent participation in similar studies. Redness is induced using 50% Glycolic Acid on the entire face and tape stripping on both forearms.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese female whose age range from 18 to 60 years old;
2. Be in general good health and good mental state;
3. Have no any broken,scars,birthmarks and other imperfections on the test area;
4. Redness/erythema≥grade 2 after modelling inducing and the score of redness must be increased after inducing;
5. Not currently be participating in any other study involving the test area(Face and Forearm);
6. Not have participated in any other study involving the test area in the past one month;
7. Be willing to read,understand and able to sign the Informed Consent Form and Photo Release From;
8. Be willing to comply with all study protocol requirements.

Exclusion Criteria:

1. Intending to get pregnant, be pregnant, be lactating, be within 6 months of delivery or be unwilling to take necessary precautions to avoid a pregnancy;
2. Having used antihistamine drugs in the past 1 week or immunosuppressants in the past 1 month;
3. Taken anti-allergic drug/injections in the past 1 month;
4. Presently have allergies, allergic dermatitis or skin disease;
5. Have sensitivity or even allergy to topical products, ingredients or fragranced products;
6. Have history of allergies;
7. Have history of suffering from skin diseases (such as psoriasis, eczema, skin cancer, etc.);
8. Have used any anti-inflammatory treatment on the test area within 2 months prior to this study starting date;
9. Has a chronic medical condition that may interfere with testing (e.g., asthma, insulin-dependent diabetes, lupus, rheumatoid arthritis or other immune/auto-immune diseases);
10. Have used any scrubs or peeling product (regardless of method) or self-tanning products or oil control products in the past 3 days;
11. Have received cosmetic medical procedures on the face (such as injectable anti-wrinkle products, cosmetic surgery, tattoo removal, home light facial procedures or home use medical devices, etc.) in the past 1 month;
12. Have excessive sun exposure or ultraviolet light exposure in the past 1 month;
13. Have applied ortho-hydroxybenzoic acid, hydroquinone in the past 3 months; or used prescriptions (such as antibiotic, retinoids, alpha hydroxyl acid and steroid), oral contraceptives；
14. Avoid providing emergency contact;
15. Subjects that are not compliant with the selection criteria or not proper for participation as determined by Principal Investigator;
16. An employee of the cosmetic companies or Shanghai China-Norm Quality technical service Co., Ltd.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Skin Erythema Index via Mexameter® MX 18 | From Baseline to 24-hour after product repeat application
Colorimetry (avalue) via Chromameter CM26dG * | from Baseline to 24-hour after product repeat application
Skin Scaliness (Desquamation) via Squamescan® 850A | from Baseline to 24-hour after product repeat application
Forearm Skin Redness (avalue) via Cross-Polarized Light Imaging * | From Baseline to 24-hour after product repeat application
  The a*value is a parameter in the CIELAB color space (also known as Lab) that quantifies a color's position along the red-green axis .
Facial Skin Redness and Colorimetry (a* value) via VISIA-CRP Imaging | from Baseline to 24-hour after product repeat application
Skin Surface Evenness (SEsc) via UV Video Capture and SELS Analysis | from Baseline to 24-hour after product repeat application

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai China-norm Quality Technical Service Co., Ltd., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided